CLINICAL TRIAL: NCT05472441
Title: Linking Education, Produce Provision, and Community Referrals to Improve Diabetes Care (LINK)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joshua Joseph, MD, Associate Professor of Medicine, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2022H0045; R01DK132403 (NIH)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Nutrition Poor; Food Deprivation
Keywords: Food Insecurity; Social Determinants of Health; Non-medical, health related social needs; Diabetes Self-Management Education and Support
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Malnutrition | interventions — Cooking

STUDY DESIGN:
Intervention Model Description: The LINK pragmatic randomized controlled trial (pRCT) uses a 2x2 factorial design to prospectively enroll study participants with type 2 diabetes and food insecurity into one of four study arms. The four study arms are: 1) Mid-Ohio Farmacy (receiving weekly produce through a consortium of local food banks); 2) Mid-Ohio Farmacy + Cooking for Diabetes (Cooking for Diabetes is a 6-week diabetes and culinary education intervention); 3) Mid-Ohio Farmacy + Health Impact Ohio Pathways Hub (The Pathways Hub uses a community health worker model to meet with participants, evaluate and address non-medical, health-related social needs); and 4) Mid-Ohio Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub).
  Participants will be randomized using a 1:1:1:1 stratified randomization scheme built into Research Electronic Data Capture (REDCap) at the participant level.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mid Ohio Food Farmacy (Active Comparator): The Food Farmacy arm receives weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective.
  Interventions: Behavioral: Mid-Ohio Food Farmacy
- Mid-Ohio Food Farmacy + Cooking for Diabetes (Experimental): The Food Farmacy + Cooking for Diabetes Arm receives weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective and Cooking for Diabetes, a 6-week diabetes self-management education and support and culinary education intervention.
  Interventions: Behavioral: Mid-Ohio Food Farmacy + Cooking for Diabetes
- Mid-Ohio Food Farmacy + Health Impact Ohio Pathways Hub (Experimental): The Food Farmacy + Health Impact Ohio Pathways Hub Arm receives weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective and has social needs address through a community health worker model at the direction of Health Impact Ohio. The community health worker meets with participants, evaluates and addresses non-medical, health-related social needs.
  Interventions: Behavioral: Mid-Ohio Food Farmacy + Health Impact Ohio Pathways Hub
- Mid-Ohio Food Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub (Experimental): The Food Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub Arm receives all 3 interventions. Participants receive weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective, Cooking for Diabetes, a 6-week diabetes self-management education and support and culinary education intervention and has social needs addressed through a community health worker model at the direction of Health Impact Ohio. The community health worker meets with participants, evaluates and addresses non-medical, health-related social needs.
  Interventions: Behavioral: Mid-Ohio Food Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub

INTERVENTIONS:
Behavioral: Mid-Ohio Food Farmacy — The Food Farmacy arm receives weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective.
  Arms: Mid Ohio Food Farmacy
Behavioral: Mid-Ohio Food Farmacy + Cooking for Diabetes — The Food Farmacy + Cooking for Diabetes Arm receives weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective and Cooking for Diabetes, a 6-week diabetes self-management education and support and culinary education intervention.
  Arms: Mid-Ohio Food Farmacy + Cooking for Diabetes
Behavioral: Mid-Ohio Food Farmacy + Health Impact Ohio Pathways Hub — The Food Farmacy + Health Impact Ohio Pathways Hub Arm receives weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective and has social needs address through a community health worker model at the direction of Health Impact Ohio. The community health worker meets with participants, evaluates and addresses non-medical, health-related social needs.
  Arms: Mid-Ohio Food Farmacy + Health Impact Ohio Pathways Hub
Behavioral: Mid-Ohio Food Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub — The Food Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub Arm receives all 3 interventions. Participants receive weekly produce through a consortium of local food banks at the direction of the Mid-Ohio Food Collective, Cooking for Diabetes, a 6-week diabetes self-management education and support and culinary education intervention and has social needs addressed through a community health worker model at the direction of Health Impact Ohio. The community health worker meets with participants, evaluates and addresses non-medical, health-related social needs.
  Arms: Mid-Ohio Food Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub

SUMMARY:
This is a pragmatic randomized controlled trial (pRCT) that aims to test the effect of produce provision, diabetes education, and community referrals on hemoglobin A1c levels in individuals with type 2 diabetes experiencing food insecurity.

DETAILED DESCRIPTION:
LINK (Linking Education, Produce Provision, and Community Referrals to Improve Diabetes Care is a 6-month pragmatic randomized controlled trial (pRCT) using a 2x2 factorial design to prospectively enroll study participants with type 2 diabetes and food insecurity into one of four study arms. The four study arms are: 1) Mid-Ohio Farmacy (receiving weekly produce through a consortium of local food banks); 2) Mid-Ohio Farmacy + Cooking for Diabetes (Cooking for Diabetes is a 6-week diabetes and culinary education intervention); 3) Mid-Ohio Farmacy + Health Impact Ohio Pathways Hub (The Pathways Hub uses a community health worker model to meet with participants, evaluate and address non-medical, health-related social needs); and 4) Mid-Ohio Farmacy + Cooking for Diabetes + Health Impact Ohio Pathways Hub). Participants will be enter

Participants will be randomized using a 1:1:1:1 stratified randomization scheme built into Research Electronic Data Capture (REDCap) at the participant level.

Primary and secondary outcomes will be collected at baseline, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes based on American Diabetes Association Criteria
* Hemoglobin A1c ≥ 7.5%
* Screen Positive on 2-item Food Security Screener

Exclusion Criteria:

* Unwilling to Attest to Release of Information to Mid-Ohio Food Collective

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 3 months
  measures average blood sugar levels over the past 3 months

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | 6 months
  measures average blood sugar levels over the past 3 months
Change in diabetes self-efficacy assessed by the Diabetes Self-Efficacy Scale | 3 months
  Diabetes self-efficacy measured via the diabetes self-efficacy scale. The Diabetes Self-Efficacy Scale has a minimum score of 10 and a maximum score of 80. A higher score indicates higher diabetes self-efficacy.
Change in diabetes self-efficacy assessed by the Diabetes Self-Efficacy Scale | 6 months
  Diabetes self-efficacy measured via the diabetes self-efficacy scale. The Diabetes Self-Efficacy Scale has a minimum score of 10 and a maximum score of 80. A higher score indicates higher diabetes self-efficacy.
Change in food security assessed using the 18-item U.S. Household Food Security Survey Module | 3 months
  Food security will be assessed using the 18-item U.S. Household Food Security Survey Module.
  For households with one or more children:
  * Raw score zero-High food security
  * Raw score 1-2-Marginal food security
  * Raw score 3-7-Low food security
  * Raw score 8-18-Very low food security
  For households with no child present:
  * Raw score zero-High food security
  * Raw score 1-2-Marginal food security
  * Raw score 3-5-Low food security
  * Raw score 6-10-Very low food security
Change in food security assessed using the 18-item U.S. Household Food Security Survey Module | 6 months
  Food security will be assessed using the 18-item U.S. Household Food Security Survey Module.
  For households with one or more children:
  * Raw score zero-High food security
  * Raw score 1-2-Marginal food security
  * Raw score 3-7-Low food security
  * Raw score 8-18-Very low food security
  For households with no child present:
  * Raw score zero-High food security
  * Raw score 1-2-Marginal food security
  * Raw score 3-5-Low food security
  * Raw score 6-10-Very low food security

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Joseph, MD, MPH, Principal Investigator — Ohio State University; Daniel Walker, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to the public as immediately and broadly as possible while safeguarding the privacy of participants and protecting confidential and proprietary data. All research data will be shared as requested in accordance with federal regulations, the Freedom of Information Act (FOIA). Requests from researchers will be reviewed by the project investigators, and we will provide the requesting researcher with the minimum necessary data; the shared data will not have any individual participant identifiers or specific clinic identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available to the public as immediately and broadly as possible while safeguarding the privacy of participants and protecting confidential and proprietary data.
Access Criteria: Requests will be reviewed by the project investigators (PI). In accordance with NIH policies and procedures regarding data use and data sharing, user registration will be required to access the files. Users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistributions of the data to third parties, and proper acknowledgement of the data resource. Any presentations, abstracts, or publications must include an acknowledgement/reference of the LINK research team.
  The requesting researcher(s) will be notified that they may only use the data for the purposes for which the data were requested and only by the individuals listed in the request. The requesting researcher(s) will be responsible for notifying the PI upon completion of analysis indicating the way the data were destroyed.

REFERENCES:
- [Derived] Walker DM, Garner JA, Hefner JL, Headings A, Jonas DE, Clark A, Bose-Brill S, Nawaz S, Seiber E, McAlearney AS, Brock G, Zhao S, Reopell L, Coovert N, Shrodes JC, Spees CK, Sieck CJ, Di Tosto G, DePuccio MJ, Williams A, Hoseus J, Baker C, Brown MM, Joseph JJ. Rationale and design of the linking education, produce provision, and community referrals to improve diabetes care (LINK) study. Contemp Clin Trials. 2023 Jul;130:107212. doi: 10.1016/j.cct.2023.107212. Epub 2023 Apr 28. PMID 37121390